CLINICAL TRIAL: NCT03085615
Title: Feeding the Critically Ill During Phases of Altered Redox Status (FEDOX): a Prospective Randomized Trial
Brief Title: Feeding the Critically Ill During Phases of Altered Redox Status
Acronym: FEDOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: American Society for Parenteral and Enteral Nutrition (Other); Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Liam McKeever, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FEDOX
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Acute Respiratory Distress Syndrome; Oxidative Stress; Euthyroid Sick Syndromes; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Euthyroid Sick Syndromes; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive either 25-30 kcals/kg or 12-14 kcals/kg. They will be followed for a maximum of 7 days or until ICU discharge. Blood draws will occur twice daily.
Who Masked: Outcomes Assessor
Masking Description: Only our lab technicians will be truly blinding to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100%NRG (Experimental): Patient will receive the enteral nutrition product Jevity 1.5 starting at 20mL per hour and increasing by 20mL every four hours until a goal rate delivering 25-30kcals/kg is achieved. If feeding is interrupted, flow rate will be adjusted to compensate for nutritional loss.
  Interventions: Other: Jevity 1.5
- 40%NRG (Active Comparator): Patient will receive the enteral nutrition product Jevity 1.5 starting at 20mL per hour and increasing by 20mL every four hours until a goal rate delivering 12-14 kcals/kg is achieved. If feeding is interrupted, flow rate will be adjusted to compensate for nutritional loss.
  Interventions: Other: Jevity 1.5

INTERVENTIONS:
Other: Jevity 1.5 — Jevity 1.5 is an enteral nutrition product delivering 1.5 kcals/mL and 0.06 g protein/mL.

SUMMARY:
The FEDOX trial is a prospective randomized clinical trial exploring oxidative stress as a mechanism of harm to explain the negative outcomes found in feeding trials that achieved caloric exposure commensurate with the nationally recommended guidelines. Due to its impact on energy metabolism, we will also explore low T3 syndrome's relationship to this mechanism. Finally, we will explore circadian patterns of diurnal/nocturnal TSH fluctuation as a potential biomarker to indicate this mechanism of harm has subsided.

This 7-day prospective randomized clinical trial is designed to address the following specific aims (SA) in ICU patients (n=40) with systemic inflammatory response syndrome.

SA1) Determine whether provision of enteral nutrition (EN) at 100% of levels in Nationally Recommended Guidelines NRG (25-30 kcals/kg, 100%NRG) early in critical illness increases reactive oxygen species (ROS) production compared to EN at 40% of NRG levels (10-12 kcals/kg, 40%NRG). Subjects will be fasted overnight and randomized to receive either 100% NRG or 40%NRG for 7 days. Plasma F2-isoprostanes will be measured daily and compared between groups through repeated measures analysis.

SA2) Determine if EN at 100%NRG interrupts the critical illness induced low T3 syndrome and subsequently further increases the ROS production compared to 40%NRG. Serum thyroid parameters (T3, T4, rT3, TSH) with be measured daily and compared between groups as above.

Mediation analysis will be used to determine the proportion of the effect of nutrition group on F2-isoprostane production explained by each thyroid parameter.

SA3) Determine if the return of diurnal/noctural fluctuations in TSH is associated with decreased nutrition-induced ROS production. Plasma TSH will be measured twice per day at 0300 and 1800hrs to determine TSH fluctuation. The interaction effect between TSH fluctuation and nutrition group on F2-isoprostane production will be assessed through repeated measures analysis. This study provides vital mechanistic insight into the impact of feeding on oxidative stress during the first week of critical illness, represents an important first step in determining the safest timing and dosage of nutrition support, and sets the foundation for future larger clinical trials on these topics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) admitted to RUMC MICU who are able to receive EN, who have two consecutive white blood cell lab values above 12,000/mm^3 or below 4,000/mm^3 plus at least one of the following 3 criteria met for at the past 12 hours will be eligible for participation. Criteria: (1) a respiratory rate greater than 20 breaths per minute or PaCO2 less than 32mmHg, (2) a heart rate greater than 90 beats per minute, or (3) a temperature greater than 100.4F or less than 96.8F.

Exclusion Criteria: Patients will be excluded if the are pregnant, have documented neurologic disease prior to admission that interferes with the capacity to give informed consent or do not require EN for their nutritional care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-10-13 (Actual)

PRIMARY OUTCOMES:
Daily Plasma F2-Isoprostane levels | 7 days
  Plasma maximum concentration of F2-isoprostanes will be quantified through liquid chromatography tandem mass spectrometry (LC-MS/MS) of plasma using a Q-trap mass spectrometer.

SECONDARY OUTCOMES:
Thyroid Stimulating Hormone (TSH) | 7 days
  TSH will be measured twice per day using commercially available immuno-assay kits.
Triiodothyronine (T3) | 7 days
  T3 will be measured daily using commercially available immuno-assay kits.
Thyroxine (T4) | 7 days
  T4 will be measured daily using commercially available immuno-assay kits.
Reverse Triiodothyronine (rT3) | 7 days
  rT3 will be measured daily using commercially available immuno-assay kits.

CONTACTS AND LOCATIONS:
Overall Officials: Liam B McKeever, MS, PhD(c), Principal Investigator — University of Illinois at Chicago; Carol A Braunschweig, PhD, Study Director — Uinversity of Illinois at Chicago; Omar Lateef, DO, Study Chair — Rush University Medical Center; Marcelo Bonini, PhD, Study Chair — University of Illinois at Chicago; Antonio Bianco, MD, PhD, Study Chair — Rush University Medical Center; Sarah J Peterson, PhD, Study Chair — Rush University Medical Center; Alan Diamond, PhD, Study Chair — University of Illinois at Chicago; Sally Freels, PhD, Study Chair — University of Illinois at Chicago
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McKeever L, Peterson SJ, Cienfuegos S, Rizzie J, Lateef O, Freels S, Braunschweig CA. Real-Time Energy Exposure Is Associated With Increased Oxidative Stress Among Feeding-Tolerant Critically Ill Patients: Results From the FEDOX Trial. JPEN J Parenter Enteral Nutr. 2020 Nov;44(8):1484-1491. doi: 10.1002/jpen.1776. Epub 2020 Jan 29. PMID 31995239
- [Derived] McKeever L, Peterson SJ, Lateef O, Freels S, Fonseca TL, Bocco BMLC, Fernandes GW, Roehl K, Nowak K, Mozer M, Bianco AC, Braunschweig CA. Higher Caloric Exposure in Critically Ill Patients Transiently Accelerates Thyroid Hormone Activation. J Clin Endocrinol Metab. 2020 Feb 1;105(2):523-33. doi: 10.1210/clinem/dgz077. PMID 31581295